CLINICAL TRIAL: NCT04972786
Title: Noninvasive Modulation of Motivational Brain Regions in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Jeremy Hogeveen, Assistant Professor, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20-623
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-06

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Sham versus active rTMS to dACC
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Magventure rTMS device enables double blinding. Participant group assignment will be blind to the participant, investigator, and outcomes assessor until all subject data has been collected, at which point the group assignment will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sham rTMS (Sham Comparator): Participants will receive sham rTMS for 10-20 minutes.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Active rTMS (Active Comparator): Participants will receive active rTMS for 10-20 minutes.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — TMS pulses will be delivered through an air-cooled coil in either a figure-eight or double-cone shape, with the latter being particularly useful for targeting deeper structures such as dACC. The first phase of the TMS protocol will involve a standardized motor-thresholding procedure, wherein peripheral responses evoked by single TMS pulses are recorded via an electromyographic recording device. In this phase, the TMS coil's stimulation intensity is titrated to a level that is comfortable yet effective at reliably exciting neuronal populations orthogonal to the coil (50% motor-evoked potentials ≥50 microvolts; typical duration≈20-40 mins). Then repetitive TMS (rTMS) will be administered to a pre-determined cortical target based on the individual's pre-TMS fMRI scan using a Localite Neuronavigation system (duration≈10-20 mins). The rTMS protocol will involve the delivery of a train of TMS pulses over a cortical target prior to performance of behavioral tasks during a post-rTMS fMRI scan.

SUMMARY:
21 healthy control participants will be recruited. On Day 1 they will complete reward-guided decision making tasks and questionnaires followed by a functional magnetic resonance imaging (fMRI) scan. On Days 2 and 3 they will receive repetitive transcranial magnetic stimulation (rTMS) targeting a specific part of the brain called the dorsal anterior cingulate cortex (dACC) or sham stimulation, and will then repeat a subset of the same decision making tasks and fMRI sequences. If brain stimulation modifies decision making and dACC activity, it could represent a novel way of treating patients with neural circuit deficits that impede motivated behavior. Of particular relevance to the current trial, this rTMS study will run in parallel with a study of apathy (i.e., diminished motivation) in patients with traumatic brain injury (TBI), with the goal of eventually leading to a patient-centered trial of rTMS treatment for this disruptive neuropsychiatric symptom.

DETAILED DESCRIPTION:
TBI is a common and impairing acquired neurological disorder caused by a concussive event to the head. Psychiatric disorders associated with impaired decision making-in particular: apathy, or diminished motivated behavior-are common post-injury in TBI. Despite the critical importance of diagnosing and characterizing psychiatric problems such as apathy in TBI, very little is known about the neuropathologies underlying apathy in this patient group.

Reinforcement learning (RL)-i.e. the process of learning the reward value of stimuli and actions-represents a fundamental cross-species construct underlying motivated decision making. Further, aberrant reward processing has been strongly implicated in symptoms of apathy in the field of computational psychiatry. Despite extensive evidence that brain injuries can lead to maladaptive motivated decision making, the specific RL aberrations that might underlie this phenomenon, and their association with psychiatric sequelae remain unclear. Therefore, extant work has failed to provide insight into the computational mechanisms underlying maladaptive decision making in patients with TBI, and such work will be critical to build a better understanding of the neuropathologies that underlie apathy in TBI. This gap in current knowledge is being targeted by a related study from which healthy controls will be recruited for the current rTMS trial.

However, even if we gain a better understanding of the RL neural mechanisms that cause aberrant motivated behavior and psychiatric sequelae in TBI, translating this into an actionable target for clinical intervention remains unclear. Psychological interventions including Cognitive-Behavioral Therapy (CBT) and Motivational Interviewing (MI) have been investigated for treating symptoms of TBI. However, the potential benefit of both CBT and MI is limited in TBI, as they both rely heavily on high-level cognitive abilities-e.g. selective attention, executive control, and metacognition/insight-that are commonly impaired in this population. In addition to psychotherapies, two categories of pharmacotherapy have been investigated to reduce psychiatric sequelae in TBI: selective serotonin reuptake inhibitors (SSRIs) and dopamine agonists. A randomized controlled trial of SSRIs for TBI failed to demonstrate reductions in patient neuropsychiatric symptoms after a 10-week intervention. Multiple pilot studies (Ns=10-11) of dopamine agonists for TBI have been conducted, demonstrating preliminary support that they may reduce apathy. Yet, a recent meta-analysis suggested a high degree of unreliability in the literature on dopamine agonism in TBI. Dopamine agonists also carry the risk of significant side effects including increased apathy or maladaptive impulsivity. Unreliability and maladaptive side effects of dopaminergic medications are likely driven by their lack of circuit-specificity: They modulate dopaminergic tone throughout the brain, rather than within a dedicated neural circuit underlying a specific symptom profile. Therefore, a more effective approach to treating apathy in TBI may involve both i) avoiding therapies that rely on high-level cognition, and ii) establishing circuit-specific approaches for ameliorating patient apathy. Precise fMRI-guided rTMS represents one possible approach. The current project aims to test the efficacy of fMRI-guided TMS to RL neural circuits anchored in dorsal anterior cingulate cortex (dACC) on motivated decision making in healthy controls. Ultimately, the hope is that this approach might represent a first step towards a potential clinical intervention for TBI patients with clinical apathy.

ELIGIBILITY:
Inclusion Criteria:

* 12 or more years of education
* ability to provide informed consent independently

Exclusion Criteria:

* Non-fluency in English
* Prior history of seizure
* contraindications to MRI (metal in the body)
* history of substance abuse (excluding moderate alcohol/cannabis usage)
* medical diagnosis of psychosis or mania

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Hogeveen, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Domenici Hall, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of participants from the local Albuquerque NM community began on 8/1/21 and ended on 6/21/23. Please note that a significant number of recruited participants attended our first baseline fMRI session but did not return for the followup rTMS intervention visits. This includes a participant that completed their baseline visit on 6/21/2023 but did not return for followup due to scheduling conflicts. In total, N=12 participants completed the intervention.
Groups:
- Active rTMS First, Then Sham rTMS: Participants first complete a Baseline Visit to identify a neural target for rTMS. Then, on Visit 2 participants receive active rTMS for 10-20 minutes prior to collection of outcome measures via fMRI. Lastly, on Visit 3, participants receive sham rTMS for 10-20 minutes, and the same outcome measures are collected.
  Repetitive Transcranial Magnetic Stimulation (rTMS): TMS pulses will be delivered through an air-cooled coil in either a figure-eight or double-cone shape, with the latter being particularly useful for targeting deeper structures such as dACC. The first phase of the TMS protocol will involve a standardized motor-thresholding procedure, wherein peripheral responses evoked by single TMS pulses are recorded via an electromyographic recording device. In this phase, the TMS coil's stimulation intensity is titrated to a level that is comfortable yet effective at reliably exciting neuronal populations orthogonal to the coil (50% motor-evoked potentials ≥50 microvolts; typical duration≈20-40 mins). Then repetitive TMS (rTMS) will be administered to a pre-determined cortical target based on the individual's pre-TMS fMRI scan using a Localite Neuronavigation system (duration≈10-20 mins). The rTMS protocol will involve the delivery of a train of TMS pulses over a cortical target prior to performance of behavioral tasks during a post-rTMS fMRI scan.
- Sham rTMS First, Then Active rTMS.: Participants first complete a Baseline Visit to identify a neural target for rTMS. Then, on Visit 2 participants receive sham rTMS for 10-20 minutes prior to collection of outcome measures via fMRI. Lastly, on Visit 3, participants receive active rTMS for 10-20 minutes, and the same outcome measures are collected.
  Repetitive Transcranial Magnetic Stimulation (rTMS): TMS pulses will be delivered through an air-cooled coil in either a figure-eight or double-cone shape, with the latter being particularly useful for targeting deeper structures such as dACC. The first phase of the TMS protocol will involve a standardized motor-thresholding procedure, wherein peripheral responses evoked by single TMS pulses are recorded via an electromyographic recording device. In this phase, the TMS coil's stimulation intensity is titrated to a level that is comfortable yet effective at reliably exciting neuronal populations orthogonal to the coil (50% motor-evoked potentials ≥50 microvolts; typical duration≈20-40 mins). Then repetitive TMS (rTMS) will be administered to a pre-determined cortical target based on the individual's pre-TMS fMRI scan using a Localite Neuronavigation system (duration≈10-20 mins). The rTMS protocol will involve the delivery of a train of TMS pulses over a cortical target prior to performance of behavioral tasks during a post-rTMS fMRI scan.
Period: Baseline MRI Scan (1 Day)
Arm/Group | Active rTMS First, Then Sham rTMS | Sham rTMS First, Then Active rTMS.
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0
Period: First Intervention (1 Day)
Arm/Group | Active rTMS First, Then Sham rTMS | Sham rTMS First, Then Active rTMS.
Started | 8 | 5
Completed | 7 | 5
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout (7 or More Days)
Arm/Group | Active rTMS First, Then Sham rTMS | Sham rTMS First, Then Active rTMS.
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Active rTMS First, Then Sham rTMS | Sham rTMS First, Then Active rTMS.
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy, non-brain-injured adult participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS First, Then Sham rTMS | Sham rTMS First, Then Active rTMS | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.14 (9.67) | 28.14 (9.67) | 28.14 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 9 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 9 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21
Immediate Expected Value (IEV) [Mean (Standard Deviation); unit: beta coefficient] — A normative computational model (POMDP) is run to fit behavioral performance on a 3-armed bandit reinforcement learning task. Weighting of immediate expected value (IEV) on this model can be generated for each subject, indicating the degree to which they relied on immediate value to drive their decisions. This between-subjects IEV parameter reflects a standardized coefficient from a multinomial logistic regression (softmax) model. Higher values on this parameter reflect a greater tendency to make decisions based on IEV.
  beta coefficient | 1.27 (0.75) | 1.34 (1.10) | 1.30 (0.93)
Effort-Based Discounting [Mean (Standard Deviation); unit: beta coefficient] — Participants make a series of effort - value tradeoff decisions on our Effort-Based Decision-Making task. Values reflect a standardized coefficient of the random subject-level intercept from a hierarchical logistic regression model fit with an interaction term, between effort and value, to index "effort-based discounting" of reward (i.e., the degree to which increases in effort level change the motivational salience of reward value on decisions). Higher values on this parameter reflect a greater tendency to de-value rewards based on increasing effort.
  beta coefficient | 0.15 (1.08) | 0.13 (1.43) | 0.14 (1.26)
dACC BOLD signal [Mean (Standard Deviation); unit: Percentage of BOLD signal change] — Encoding of trial-by-trial immediate expected value (IEV) in dorsal anterior cingulate cortex (dACC) region-of-interest that was targeted with rTMS. Expressed in units of BOLD % signal change.
  Percentage of BOLD signal change | -1.39 (1.26) | -0.92 (1.12) | -1.16 (1.19)

OUTCOME MEASURES:

1. Primary Outcome: dACC BOLD Signal (After Active rTMS Session)
Description: Encoding of trial-by-trial immediate expected value (IEV) in dorsal anterior cingulate cortex (dACC) region-of-interest that was targeted with rTMS. Expressed in units of BOLD % signal change. This primary outcome reflects IEV encoding in this region immediately after active rTMS.
Time Frame: 30 minutes post-rTMS
Population: Several participants came for baseline visit but did not return for rTMS visits. Once participant from Arm 1 elected to discontinue rTMS and did not return for their sham visit.
Measure: Mean (Standard Deviation); unit: Percentage of BOLD signal change
Arm/Group | Active rTMS First, Then Sham rTMS | Sham rTMS First, Then Active rTMS
Number analyzed (Participants) | 8 | 5
Percentage of BOLD signal change | -1.14 (0.92) | -1.27 (0.91)

2. Primary Outcome: Immediate Expected Value (IEV; After Active rTMS Visit)
Description: A normative computational model (POMDP) is run to fit behavioral performance on a 3-armed bandit reinforcement learning task. Weighting of immediate expected value (IEV) on this model can be generated for each subject, indicating the degree to which they relied on immediate value to drive their decisions. This between-subjects IEV parameter reflects a standardized coefficient from a multinomial logistic regression (softmax) model. Higher values indicate a greater tendency to rely on IEV when making choices.
Time Frame: 30 minutes post-rTMS
Population: Several participants completed baseline visit but did not return for rTMS visits.
Measure: Mean (Standard Deviation); unit: beta coefficient
Groups:
- Sham rTMS First, Then Active rTMS: Participants first complete a Baseline Visit to identify a neural target for rTMS. Then, on Visit 2 participants receive active rTMS for 10-20 minutes prior to collection of outcome measures via fMRI. Lastly, on Visit 3, participants receive sham rTMS for 10-20 minutes, and the same outcome measures are collected.
  Repetitive Transcranial Magnetic Stimulation (rTMS): TMS pulses will be delivered through an air-cooled coil in either a figure-eight or double-cone shape, with the latter being particularly useful for targeting deeper structures such as dACC. The first phase of the TMS protocol will involve a standardized motor-thresholding procedure, wherein peripheral responses evoked by single TMS pulses are recorded via an electromyographic recording device. In this phase, the TMS coil's stimulation intensity is titrated to a level that is comfortable yet effective at reliably exciting neuronal populations orthogonal to the coil (50% motor-evoked potentials ≥50 microvolts; typical duration≈20-40 mins). Then repetitive TMS (rTMS) will be administered to a pre-determined cortical target based on the individual's pre-TMS fMRI scan using a Localite Neuronavigation system (duration≈10-20 mins). The rTMS protocol will involve the delivery of a train of TMS pulses over a cortical target prior to performance of behavioral tasks during a post-rTMS fMRI scan.
Arm/Group | Active rTMS First, Then Sham rTMS | Sham rTMS First, Then Active rTMS
Number analyzed (Participants) | 8 | 5
beta coefficient | 1.22 (0.76) | 1.62 (0.87)

3. Primary Outcome: Effort-Based Discounting (After Active rTMS)
Description: Participants make a series of effort - value tradeoff decisions on our Effort-Based Decision-Making task. Values reflect a standardized coefficient of the random subject-level intercept from a hierarchical logistic regression model fit with an interaction term, between effort and value, to index "effort-based discounting" of reward (i.e., the degree to which increases in effort level change the motivational salience of reward value on decisions). Higher values indicate a greater tendency to de-value rewards based on increasing effort level.
Time Frame: 30 minutes post-rTMS
Population: Several participants did the baseline visit but did not return to complete the rTMS visits.
Measure: Mean (Standard Deviation); unit: beta coefficient
Groups:
- Active rTMS First, Then Sham rTMS: Participants will receive sham rTMS for 10-20 minutes.
  Repetitive Transcranial Magnetic Stimulation: TMS pulses will be delivered through an air-cooled coil in either a figure-eight or double-cone shape, with the latter being particularly useful for targeting deeper structures such as dACC. The first phase of the TMS protocol will involve a standardized motor-thresholding procedure, wherein peripheral responses evoked by single TMS pulses are recorded via an electromyographic recording device. In this phase, the TMS coil's stimulation intensity is titrated to a level that is comfortable yet effective at reliably exciting neuronal populations orthogonal to the coil (50% motor-evoked potentials ≥50 microvolts; typical duration≈20-40 mins). Then repetitive TMS (rTMS) will be administered to a pre-determined cortical target based on the individual's pre-TMS fMRI scan using a Localite Neuronavigation system (duration≈10-20 mins). The rTMS protocol will involve the delivery of a train of TMS pulses over a cortical target prior to performance of behavioral tasks during a post-rTMS fMRI scan.
- Sham rTMS First, Then Active rTMS: Participants will receive active rTMS for 10-20 minutes.
  Repetitive Transcranial Magnetic Stimulation: TMS pulses will be delivered through an air-cooled coil in either a figure-eight or double-cone shape, with the latter being particularly useful for targeting deeper structures such as dACC. The first phase of the TMS protocol will involve a standardized motor-thresholding procedure, wherein peripheral responses evoked by single TMS pulses are recorded via an electromyographic recording device. In this phase, the TMS coil's stimulation intensity is titrated to a level that is comfortable yet effective at reliably exciting neuronal populations orthogonal to the coil (50% motor-evoked potentials ≥50 microvolts; typical duration≈20-40 mins). Then repetitive TMS (rTMS) will be administered to a pre-determined cortical target based on the individual's pre-TMS fMRI scan using a Localite Neuronavigation system (duration≈10-20 mins). The rTMS protocol will involve the delivery of a train of TMS pulses over a cortical target prior to performance of behavioral tasks during a post-rTMS fMRI scan.
Arm/Group | Active rTMS First, Then Sham rTMS | Sham rTMS First, Then Active rTMS
Number analyzed (Participants) | 8 | 5
beta coefficient | 0.35 (1.01) | -0.62 (0.65)

4. Primary Outcome: dACC BOLD Signal (After Sham rTMS Session)
Description: Encoding of trial-by-trial immediate expected value (IEV) in dorsal anterior cingulate cortex (dACC) region-of-interest that was targeted with rTMS. Expressed in units of BOLD % signal change. This primary outcome reflects IEV encoding in this region immediately after sham rTMS.
Time Frame: 30 minutes post-rTMS
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of BOLD signal change
Arm/Group | Active rTMS First, Then Sham rTMS | Sham rTMS First, Then Active rTMS
Number analyzed (Participants) | 8 | 5
Percentage of BOLD signal change | -1.18 (1.61) | -0.96 (0.94)

5. Primary Outcome: Immediate Expected Value (IEV; After Sham rTMS Visit)
Description: as for outcome 2
Time Frame: 30 minutes post-rTMS
Population: Several participants completed baseline visit but did not return for rTMS visits.
Measure: Mean (Standard Deviation); unit: beta coefficient
Arm/Group | Active rTMS First, Then Sham rTMS | Sham rTMS First, Then Active rTMS
Number analyzed (Participants) | 8 | 5
beta coefficient | 1.06 (0.56) | 1.32 (1.10)

6. Primary Outcome: Effort-Based Discounting (After Sham rTMS)
Description: as for outcome 3
Time Frame: 30 minutes post-rTMS
Population: Several participants did the baseline visit but did not return to complete the rTMS visits.
Measure: Mean (Standard Deviation); unit: beta coefficient
Arm/Group | Active rTMS First, Then Sham rTMS | Sham rTMS First, Then Active rTMS
Number analyzed (Participants) | 8 | 5
beta coefficient | 0.08 (0.12) | 0.13 (0.18)

ADVERSE EVENTS:
Time Frame: The duration of time over which each participant was assessed was a median of 41.5 days across the sample of participants that completed all three study visits.
Description: Three types of adverse event data are to be reported: "All-Cause Mortality," "Serious," and "Other (Not Including Serious)" Adverse Events.
  1. All-Cause Mortality.
  2. Serious Adverse Events.
  3. Other (Not Including Serious) Adverse Events.
Groups:
- Active rTMS: Repetitive Transcranial Magnetic Stimulation (rTMS): TMS were delivered through an air-cooled coil in either a double-cone shape placed over dACC. The first phase of the TMS protocol involved a standardized motor-thresholding procedure, wherein peripheral responses evoked by single TMS pulses were recorded via an electromyographic recording device. In this phase, the TMS coil's stimulation intensity is titrated to a level that is comfortable yet effective at reliably exciting neuronal populations orthogonal to the coil (50% motor-evoked potentials ≥50 microvolts; typical duration≈20-40 mins). Then repetitive TMS (rTMS) was administered to a pre-determined cortical target based on the individual's pre-TMS fMRI scan using a Localite Neuronavigation system (duration≤10 mins). The rTMS protocol will involve the delivery of a train of TMS pulses over a cortical target prior to performance of behavioral tasks during a post-rTMS fMRI scan.
- Sham rTMS: Sham Repetitive Transcranial Magnetic Stimulation (sham rTMS): TMS were delivered through an air-cooled coil in either a double-cone shape placed over dACC. The first phase of the TMS protocol involved a standardized motor-thresholding procedure, wherein peripheral responses evoked by single TMS pulses were recorded via an electromyographic recording device. In this phase, the TMS coil's stimulation intensity is titrated to a level that is comfortable yet effective at reliably exciting neuronal populations orthogonal to the coil (50% motor-evoked potentials ≥50 microvolts; typical duration≈20-40 mins). Then repetitive TMS (rTMS) was administered to a pre-determined cortical target based on the individual's pre-TMS fMRI scan using a Localite Neuronavigation system (duration≤10 mins). The rTMS protocol will involve the delivery of a train of TMS pulses over a cortical target prior to performance of behavioral tasks during a post-rTMS fMRI scan.
  For the sham procedure, subtle tactile stimulation was applied via electrodes underneath the rTMS coil. A sham coil was used that mimicked the sound of the active rTMS delivery without modulating brain activity. This was used to mirror the sensory and placebo effects of the rTMS intervention without neuromodulation.
Arm/Group | Active rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS (N=12) | Sham rTMS (N=12)
Discomfort during Active rTMS (Product Issues) | 1 (1) | 0 (0) — During their first rTMS visit, one participant experienced sufficient facial nerve irritation during active rTMS dlivery that they were discontinued from participating in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT04972786/Prot_SAP_002.pdf
  • Informed Consent Form (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT04972786/ICF_001.pdf